CLINICAL TRIAL: NCT04735107
Title: Low Anterior Resection Combined With Transanal Reinforcement and Endoluminal Sponge Vacuum Drainage
Brief Title: Mucosal Flap Reinforced Colorectal Anastomosis and Trans-Anal Vacuum Drainage: A Feasibility Study
Acronym: Endodrain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Comenius University (Other)
Collaborators: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Alexander Ferko, Clinical professor, Comenius University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No 2018/16-UKMT-12
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Rectal Cancer
Keywords: low anterior resection; anastomotic dehiscence
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reinforcement (Experimental): Low anterior resection + mucosa flap reinforcement + vacuum sponge endoluminal drainage
  Interventions: Procedure: colorectal anastomosis reinforcement and trans-anal drainage

INTERVENTIONS:
Procedure: colorectal anastomosis reinforcement and trans-anal drainage — Circular mucosal flap created to cover stapled anastomosis + vacuum sponge drainage
  Other Names: Mucosal flap double-stapled anastomosis reinforcement

SUMMARY:
Background: Dehiscence of colorectal anastomosis is a serious complication associated with increased mortality and impaired functional and oncological outcomes. We hypothesised that anastomosis reinforcement and vacuum trans-anal drainage could eliminate some risk factors of colorectal anastomotic dehiscence,including mechanically stapled anastomosis instability and local infection.

DETAILED DESCRIPTION:
The study included consecutive patients older than 18 years who had low anterior resection of the rectum and anastomosis performed by double-stapler technique, for rectal cancer located within 10 cm from the anal verge. All patients had undergone pelvic magnetic resonance imaging. Nutrition screening was performed in all patients. If patients had undergone neoadjuvant chemoradiotherapy (CHRT), restaging was performed within 6 weeks of CHRT completion, and surgery was performed 10 weeks after CHRT completion. For the surgical procedure, low anterior resection (LAR) was performed by experienced surgeons who perform more than 50 rectal procedures per year and have sufficient expertise in minimally invasive surgery. Oral bowel preparation was used preoperatively and antibiotics were administered according to protocol.

1. Surgical technique

   The procedure milestones (descending colon blood perfusion, tension-free anastomosis, safely performed stapled anastomosis and reinforcement, and safely performed mucosal flap) were defined. Simultaneous checkpoints to control milestones were identified and methodology of their documentation (video, photography) were defined. The purpose was to achieve demonstrable control over the individual steps during the surgical procedure.

   1.1 Abdominal phase

   Laparoscopic procedures were performed in the Lloyd-Davis position, using the 4-ports technique. During the abdominal phase, dissection was guided by a medio-lateral approach. A high tie of the a. mesenterica inferior (AMI) was performed in all patients. Dissection was performed medio-laterally and down to the pelvic floor according to the principles of total mesorectal excision (TME). The rectum was transected using an endostapler after lavage with Betadine solution (Egis Pharmaceuticals, PLS, Budapest, Hungary). Furthermore, the splenic flexure was fully mobilized using a combination of medio-lateral and lateral approaches. In most cases, the inferior mesenteric vein was divided.

   The marginal artery was dissected and the character of arterial blood flow was carefully evaluated; pulsatile arterial blood flow was considered as sign of adequate colon perfusion (Checkpoint 1).

   A specimen of tumor was pulled through the minilaparotomy and resected. The descending colon was divided at the level of the distal part and the colonic mucosa was again evaluated with respect to blood perfusion; a light red or pink colored mucosa and fresh light red capillary bleeding were considered as signs of good colonic mucosa perfusion (Checkpoint 2). The colon needed to lie freely in the sacrum excavation and no tension was allowed on the mesenterial site. This was confirmed by lifting the colon ventrally from the sacrum at the promontory level after anastomosis construction (Checkpoint 3). The anastomosis was performed end-to-end using a double-stapler technique, strictly between the descending colon and rectum in a tension-free manner. A pelvic drain was left in place till the third postoperative day.

   1.2 Trans-anal phase

   As part of the trans-anal phase, a Lone Star retractor (Cooper Surgical, Inc. USA) and a plastic single use anoscope were applied. An initial, careful inspection and manual check of the stapler anastomosis integrity, the blood supply to the colonic mucosa, and signs of a tension-free anastomosis were performed (Checkpoint 4). The mucosal flap was subsequently created using individual polydiaxone (PDS) II 5/0 sutures (polydiaxonone, Ethicon, Johnson&Johnson, USA): individual stitches were placed on each quadrant; and then another four stitches were applied in between. It is important to note that the condition of the mucosal flap upon creation were signs of a floppy, prolapsing colonic wall into the anastomosis. Finally, a sponge soaked (Endo-SPONGE, B. Braun, Germany) with povidone-iodine (Betadine, Egis Pharmaceuticals, Budapest, Hungary) was introduced into the anastomosis. The trans-anal sponge drain was removed 24 hrs postoperatively.

   1.3 Fecal diversion

   The decision on diversion was based on intraoperative checkpoint adherence: when Checkpoint 6 and 7 were not fulfilled, an ileostomy was created.
2. Follow up

The data regarding the type of procedure, type of anastomosis, stapler diameter, the number of stapler cartridges used, dissection of the mesenteric blood vessels, and complete histopathology were collected prospectively. C-reactive protein (CRP) levels were assessed on the third and fifth day after surgery.0 Patients were followed up for 3 months, and postoperative endoscopy was performed before discharge, usually on postoperative day 7, 1 month after surgery, and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed extraperitoneal rectal cancer, cT1-cT4
* Patient with low anterior resection and double-stapled anastomosis technique

Exclusion Criteria:

* Patients not provided written informed consent
* Patients with cT4: with pelvic side wall involement, requiring pelvic more extensive procedure
* Patients with recurrent rectal cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of anastomotic leak | 30 days
  Leak of colorectal anastomosis proven by endoscopy/or/and computed tomography
Defunction ileostomy rate | 30 days
  Rate of fecal diversion in group of treated patients

SECONDARY OUTCOMES:
Postoperative morbidity | 30 days
  Complications in postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ferko, Prof.MD,PhD, Principal Investigator — Comenius University, Jessenius Medical Faculty in Martin
Locations (1):
- University Hospital Martin, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferko A, Vana J, Adamik M, Svec A, Zacek M, Demeter M, Grendar M. Mucosa plication reinforced colorectal anastomosis and trans-anal vacuum drainage: a pilot study with preliminary results. Updates Surg. 2021 Dec;73(6):2145-2154. doi: 10.1007/s13304-021-01105-4. Epub 2021 Jun 5. PMID 34089500